CLINICAL TRIAL: NCT07068334
Title: Effects of Functional and Kinetic Treatment With Rehabilitation (FAKTR) Therapy on Muscle Activity, Ankle Proprioception and Foot Biomechanics in Over Pronated Patients With Chronic Non-specific Low Back Pain
Brief Title: Effects of FAKTR Therapy on Muscle Activity, Ankle Proprioception and Foot Biomechanics in OP With Low Back Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PhDRSW/Batch-Fall23/2222
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Physical Therapy: (Experimental)
  Interventions: Combination Product: Traditional Physical Therapy
- Traditional Physical Therapy + FAKTR (Active Comparator)
  Interventions: Combination Product: Traditional Physical Therapy + FAKTR

INTERVENTIONS:
Combination Product: Traditional Physical Therapy — Short foot exercises. Towel-curl exercise. Heel raise exercise. Calf stretch.
  Arms: Traditional Physical Therapy:
Combination Product: Traditional Physical Therapy + FAKTR — Short foot exercises. Towel-curl exercise. Heel raise exercise. Calf stretch.
  FAKTR Functional and Kinematic Treatment with Rehabilitation) technique:
  The FAKTR (Functional and Kinematic Treatment with Rehabilitation) technique applied is a modified IASTM technique in the pain-provocative position (incorporating static positions, motions, functional movements, resistance, and proprioceptive positions).
  Arms: Traditional Physical Therapy + FAKTR

SUMMARY:
Low back pain is sometimes non-specific, leading to pain and spasm due to muscle imbalance causing changes in biomechanical properties, back and limb muscles, leading to dictating a significant association between low back pain and overpronation. FAKTR (functional and kinetic treatment with rehabilitation) Therapy employs this mobilization with proprioception and resistance treating these biomechanical changes.

DETAILED DESCRIPTION:
This study aims to determine the effects of FAKTR (functional and kinetic treatment with rehabilitation) therapy on muscle activity, ankle proprioception and foot biomechanics on over-pronated foot in patients with chronic non-specific low back pain. This study will be a Randomized Controlled trial and will be conducted on sample size of 60 patients, will be taken by consecutive sampling techniques. Patients will be randomly assigned into two groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 25-45
* Both males and females
* History of three or more occurrences of lower back pain in the year before the study. - The diagnosis is confirmed by the pain experienced between the inferior gluteal folds and the costal margins.
* Moderate to severe pain is measured using a Numerical pain rating scale.
* Foot Posture Index score higher than +6. A total score ranging from -12 to +12 is obtained by measuring the subject's six feet using the Foot Posture Index (FPI). The following are the reference values for the posture of the feet: A neutral position is indicated by 0 to +5, a pronated position by +6 to +9, a hyper-pronated position by +10 to +12, a supinated position by -1 to -5, and a very supinated position by -6 to - 12.

Exclusion Criteria:

* No recent history of lower limb fractures or injuries
* No history of surgical treatment experience for spinal stenosis, spina bifida, or disc herniation
* No neurological issues or constriction of the nerve roots.
* Previously diagnosed with Osteoporosis.
* SIJ dysfunction evaluated by Compression test positive
* Congenital deformities

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2025-04-17 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale (NPRS) | 18 Months
  This scale will be used to determine the participant's pain threshold. This scale has a 0 to 10 range. The pain scale goes from zero (no pain) to ten (highest agony). High test-retest reliability has been demonstrated using NPRS (r = 0.96 and 0.95, respectively)
Balance of the Error Scoring System (BESS) | 18 Months
  The BESS incorporates three stances-double, single, and tandem-to assess static balancing skills. It takes 20 seconds to accomplish each stance. In the BESS, a participant's score is determined by how many mistakes they make; each mistake is worth one point. Opening the eyes, stepping, stumbling, falling, staying out of position for more than five seconds, shifting the hip into more than 30 degrees of flexion or abduction, elevating the forefoot or heel, and lifting the hands of the iliac crests are all examples of potential mistakes. Each posture is permitted to have a maximum of 10 points. A contestant will receive a maximum score of 10 for that stance if they are unable to hold it for five seconds. The total score of the BESS ranges from 0 to 60 and is calculated as the sum of the error points given for each of the six stances.
Oswestry Disability Index (ODI) | 18 Months
  The Oswestry Handicap Index, also known as the Oswestry Low Back Pain Disability Questionnaire, is a very crucial instrument to assess a patient's functional disability over the long term. The evaluation is regarded as the "gold standard" for measuring low-back functional results. The final score/index is on a scale of 0 to 100. Scores range from 0 to 20 for mild impairment, 21 to 60 for severe disability, 61 to 80 for crippled, and 81 to 100 for bed bound.
Valgus angle by goniometer | 18 Months
  The hindfoot valgus angle, also known as the valgus angle behind the ankle, is calculated by drawing a line between the midline of the heel and the midline of the lower part of the leg when the participant is in prone lying. After the procedure, the participant will be instructed to stand up, and the angle will be measured once more using a goniometer. Overpronation is defined as a value greater than nine, with 180 degrees being the usual angle. The reliability for angle dorsiflexion is 0.12-0.73 ICC, and the validity is 0.51-0.83

CONTACTS AND LOCATIONS:
Locations (1):
- Arif memorial teaching hospital, ferozepur road, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No